CLINICAL TRIAL: NCT02935621
Title: Behavioral Interventions for Active Duty Service Members and Veterans With Chronic Pain Conditions and Opioid Related Problems
Brief Title: Behavioral Interventions for Active Duty Service Members and Veterans With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Garland, Ph.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00091781
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Oriented Recovery Enhancement (Experimental): Participants will attend a Mindfulness-Oriented Recovery Enhancement (MORE) group weekly for eight weeks.
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE)
- Support Group (Active Comparator): Participants will attend a support group weekly for eight weeks.
  Interventions: Behavioral: Support Group

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE) — Mindfulness-Oriented Recovery Enhancement (MORE) is a group behavioral intervention that unites mindfulness training, cognitive reappraisal, and positive psychological principles into an integrative intervention strategy targeting mechanisms of pain and opioid misuse.
  Arms: Mindfulness-Oriented Recovery Enhancement
Behavioral: Support Group — A conventional support group will allow participants to express emotions, share experiences, and receive social support under the guidance of a skilled therapist.
  Arms: Support Group

SUMMARY:
The central aim of this proposed study is to test a multimodal, mindfulness-oriented intervention designed to disrupt the risk chain leading to prescription opioid dose escalation, opioid misuse and opioid addiction, which are mounting threats to active duty service members and Veterans with chronic pain conditions, who may develop disordered opioid use as a consequence of long-term opioid pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* men/women ≥18 years of age
* ability to understand and speak the English language
* current chronic pain diagnosis (including but not limited to ICD-9 diagnoses 338.0, 338.2xx, 338.
* current use of prescription opioids for >3 consecutive months.

Exclusion Criteria:

* Mindfulness training experience (participation in MBSR/MBRP)
* opioid withdrawal evidenced by score ≥13 on the Clinical Opiate Withdrawal Scale
* current cancer diagnosis
* having a psychiatric or medical condition that precludes the ability to provide informed consent or participation in outpatient treatment (e.g., psychosis, mania, acute intoxication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in opioid misuse | Baseline, and through 6 months post-treatment
  Change in Current Opioid Misuse Measure from baseline through study completion (6 months post-treatment). Opioid misuse as evidenced by triangulated aggregate of Current Opioid Misuse Measure and/or clinician assessment via Addiction Behaviors Checklist and/or urine screen
Change in pain severity and interference | Baseline, and through 6 months post-treatment
  Change on Brief Pain Inventory items from baseline through study completion (6 months post-treatment)

SECONDARY OUTCOMES:
Change in opioid craving | Baseline, during treatment
  Change in EMA opioid craving measure from Wasan et. al 2012 from baseline through study treatment completion
Change in psychological distress | Baseline, and through 6 months post-treatment
  Change in Depression Anxiety Stress Scale from baseline through study completion (6 months post-treatment)
Change in opioid dose (in morphine equivalents) | Baseline, during treatment, and through 6 months post-treatment
  Change from baseline through study completion (6 months post-treatment)
Change in post-traumatic stress | Baseline, and through 6 months post-treatment
  Change in Post-Traumatic Stress Checklist-Military from baseline through study completion (6 months post-treatment)
Change in resilience | Baseline, and through 6 months post-treatment
  Change in Response to Stressful Events Scale from baseline through study completion (6 months post-treatment)

OTHER OUTCOMES:
Change in nonreactivity | Baseline, and through 6 months post-treatment
  Change in Five Facet Mindfulness Questionnaire nonreactivity subscale from baseline through study completion (6 months post-treatment)
Change in reinterpretation of pain sensations | Baseline, and through 6 months post-treatment
  Change in Coping Strategies Questionnaire reinterpretation of pain subscale from baseline through study completion (6 months post-treatment)
Change in emotion regulation | Baseline, post-treatment (8 weeks from beginning of treatment)
  Change from baseline through post-treatment as measured by responses on the Emotion Regulation Task.
Change in positive emotion | Baseline, and through 6 months post-treatment
  Change in Positive and Negative Affect Scale from baseline through study completion (6 months post-treatment)
Change in cue-reactivity | Baseline, post-treatment (8 weeks from beginning of treatment)
  Change from baseline through post-treatment as evidenced by attentional bias and autonomic responses during lab-based task involving rapid presentation of cues designed to measure cue-reactivity
Change in attention to positive information | Baseline, and through 6 months post-treatment
  Change in Attention to Positive and Negative Information Scale from baseline through study completion (6 months post-treatment)
Change in interoceptive awareness | Baseline, and through 6 months post-treatment
  Change in Multidimensional Assessment of Interoceptive Awareness from baseline through study completion (6 months post-treatment)
Change in EEG spectral power during mindfulness | Baseline, post-treatment (8 weeks from beginning of treatment)
  In an ancillary mechanistic sub-study, a subset of participants will be assessed with EEG during a laboratory-based mindfulness meditation practice session. EEG frequency analyses will compute spectral power bands during mindfulness.
Change in anhedonia | Baseline, and through 6 months follow-up
  Change in Snaith Hamilton Anhedonia and Pleasure Scale from baseline through 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garland, PhD, Principal Investigator — University of Utah
Locations (1):
- George Wahlen VA Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided